CLINICAL TRIAL: NCT04802538
Title: A Phase 1 Clinical Trial to Assess the Performance and Safety of a Novel Ostomy Ring (OstoRing®) to Improve Ileostomy and Colostomy Management
Brief Title: Performance and Safety of a Novel Ostomy Ring to Improve Ileostomy and Colostomy Management
Acronym: OstoRing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to terminate study due to insufficient recruitment.
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: EH19-278
Record Dates: First submitted 2021-01-25; First posted 2021-03-17 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2022-03

CONDITIONS: Stoma Site Leakage
Keywords: ileostomy; colostomy; stoma

STUDY DESIGN:
Intervention Model Description: Early feasibility device study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Group (Experimental): All patients will begin the study by using their normal ostomy pouching equipment for 28 days. This will be followed by a transition to using the OstoRing® for 28-47 days.
  Interventions: Device: OstoRing®

INTERVENTIONS:
Device: OstoRing® — Participants will use the OstoRing® along with their standard pouching equipment.

SUMMARY:
In this study, a novel ostomy ring device will be assessed for safety and efficacy in increasing the lifespan of ostomy pouching equipment.

DETAILED DESCRIPTION:
In this crossover design trial, patients will be asked to first wear their normal ostomy pouching equipment for 28 days followed by 28 days with the OstoRing®. Patients may choose to continue using the OstoRing for an additional 19 days. Study visits will occur between each section of the trial and will involve a skin assessment and quality of life questionnaires. Additionally, over the course of the trial, participants will be asked to fill out a survey and take a picture of their stoma with ostomy pouching change.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age and have full legal capacity
* Have had an end or loop ileostomy or colostomy for at least 6 months.
* Have used a Hollister 2 piece New Image pouching system for at least 8 weeks
* Able to provide informed consent
* Have a stoma with a diameter of 57mm or less
* Change their pouching system at least two times in seven days

Exclusion Criteria:

* Unable to give informed consent.
* Are pregnant or currently breastfeeding.
* In the last 2 months has received or is currently receiving, chemotherapy or radiation therapy.
* In the last month has received or is currently receiving systemic or local steroid treatment in the peristomal area.
* Currently suffering from severe peristomal skin problems such as peristomal pyoderma, abscess.
* Currently suffering from a peristomal hernia.
* Known hypersensitivity toward any of the test product (OstoRing® is made of surgical grade stainless steel)
* In the last 30 days has participated or is currently participating in a clinical study
* Assessed with an ostomy skin tool score of ≥3

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Pouching Equipment Wear Time/Lifespan | 75 days
  Mean pouching system wear time will be calculated with and without the OstoRing®.
Coloplast Tool Skin Assessment Score | 75 days
  The skin surrounding the peristomal area will be assessed at all study visits utilizing the coloplast skin score tool. Skin score may range from 0 to 15 with a smaller score indicating better skin condition in the peristomal area.

SECONDARY OUTCOMES:
City of Hope Quality of Life Ostomy Questionnaire Score | 75 days
  Quality of life will be assessed at all study visits utilizing the City of Hope Quality of Life Ostomy Questionnaire. This instrument contains 43 questions with answers on a Likert scale from 1 to 10. The final score is the sum of all responses divided by the total number questions which gives a final score from 1 to 10. Greater score on this survey is indicative of a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene F Yen, MD, MBA, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem Evanston Hospital, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT04802538/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT04802538/ICF_000.pdf